CLINICAL TRIAL: NCT02107144
Title: The Study to Assess the Effect of Trimetazidine on Index of Microcirculatory Resistance (IMR), Measured by Coronary Pressure and Temperature Wire, in Patients With Stable Coronary Artery Disease
Brief Title: The ImPact of Trimetazidine on MicrOcirculation After Stenting for Stable Coronary Artery Disease
Acronym: PATMOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Center Zemun (Other)
Responsible Party: Principal Investigator, Ivan Ilic, MD PhD, interventional cardiologist, Clinical Hospital Center Zemun
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZEM - CARD - 002
Record Dates: First submitted 2014-03-29; First posted 2014-04-08 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Microcirculation; Vascular Resistance
Keywords: trimetazidine; microcirculation; stenting; pressure wire
MeSH Terms: conditions — Coronary Artery Disease | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trimetazidin (Experimental): Patients, who are trimetazidine (TMZ) naïve, will be randomly assigned to receive trimetazidine plus previous medications (TMZ group) 48h before scheduled PCI- Paients that are TMZ naïve and randomized to TMZ group will be given oral loading of 70mg TMZ.
  Interventions: Drug: trimetazidine
- Control (No Intervention): Patients, who are TMZ naïve, will be randomly assigned to receive just previous cardiac medication (Control group).

INTERVENTIONS:
Drug: trimetazidine — After being randomized to Trimetazidin and cardiac medication vs. only cardiac medication, patient will undergo scheduled PCI of single, new, native coronary artery lesion using balloon predilatation and subsequent stenting.
  Other Names: Vastarel MR; Preductal MR; Trimetacor
  Arms: trimetazidin

SUMMARY:
The study should enrol 50 patients with stable coronary artery disease scheduled for elective percutaneous coronary intervention of single, de novo lesion of native coronary artery. Patients will be randomized to orally given trimetazidine on top of standard medical therapy for stable coronary artery disease versus standard therapy only. The randomization will begin 48 hrs before intervention. Index of microcirculatory resistance (IMR) will be measured by thermodilution method using coronary pressure and temperature wire before and after stent implantation. Echocardiography will be performed before intervention and within 30 minutes after intervention. Patients will be followed clinically for a period of one year.

DETAILED DESCRIPTION:
The study is prospective, single blinded randomized study that will be performed in a single tertiary cardiovascular centre. The inclusion criteria for the study are the presence of the stable angina or positive stress test, Canadian Cardiovascular Society (CCS) class less than IV and an indication for percutaneous intervention of a single, de novo, native coronary artery lesion with diameter stenosis greater than 70%. Exclusion criteria are left ventricular systolic function (LVEF) less than 30%, acute coronary syndrome, a history of previous myocardial infarction in the territory supplied by the treated coronary artery, existence of the collateral circulation to another coronary artery supplied by the treated vessel, chronic total occlusion, significant bifurcation lesion, previous surgical revascularization, significant renal function impairment (GFR less than 60ml/min), allergy to any constituents of trimetazidine, aspirin and antiplatelet medications used after PCI, contrast agents, contraindication to adenosine use. The patient with disorders like Parkinson disease, parkinsonian symptoms, tremors, restless leg syndrome, and other related movement disorders will also be excluded from the study.

Patients, who are trimetazidine naïve, will be randomly assigned to receive either trimetazidine plus previous medications (TMZ group) 48h before scheduled PCI or just previous medication (Control group). Paients that are TMZ naïve and randomized to TMZ group will be given loading of 70mg of TMZ on day 0. The PCI operator would not be aware if the patient receives TMZ. All patients will be pretreated before PCI with aspirin 100mg/day, Clopidogrel 75mg/day seven days before the procedure. Patient will be asked to sign informed consent form before entering the study and the study protocol was approved by Ethics committee of Clinical Hospital Center Zemun.

Patients will undergo PCI intervention on day 2. Before PCI patients will receive heparin 80 - 100 IU/kg iv. PCI procedure has to be performed with angioplasty balloon predilation of the treated lesion to avoid influence of direct stenting on IMR measurement. The stenting will be performed according to operator's preference. The fractional flow reserve (FFR), coronary flow reserve (CFR) and IMR will be measured before and after PCI using coronary pressure - / thermistor - tipped wire (Radi Pressure Wire Certus, St Jude Medical, Uppsala, Sweden). Maximal hyperemia will be achieved using iv infusion of adenosine (140mcg/kg/min) during the procedure. The pressure wire will be advanced through 6F guiding catheter to position the pressure sensor at a point 10 mm distal to the distal end of the stenosis or the stent after PCI procedure. Three injections of 3ml normal saline at room temperature will be administered via guiding catheter at baseline before starting PCI procedure and at maximal hyperemia. The transit time will be measured as the time that elapses between the moment when one-half of the saline had been injected (defined as T0, and determined on the temperature curve from the shaft of the wire) and the moment when one-half of the saline had passed the sensor. Simultaneous recordings of mean aortic pressure (guiding catheter, Pa) and mean distal coronary pressure (distal pressure sensor, Pd) will also be obtained at baseline and during maximal hyperemia. FFR will be calculated by dividing the mean distal coronary pressure (Pd) by the mean aortic pressure (Pa) during maximal hyperemia. CFR will be calculated as a ratio of mean transit time at basal condition (Tbas) and after inducing hyperemia (Thyp). The IMR will be calculated using the following equation: IMR = Pa x Thyp [(Pd - Pw) / (Pa - Pw)], where Pw is the coronary wedge pressure. Pw will be measured as the distal coronary pressure Pd (from the distal pressure and temperature sensor) during complete balloon occlusion of the vessel with the angioplasty balloon during PCI.

Coronary angiograms will be analyzed offline using a computer-assisted, automated edge-detection algorithm using dedicated software Axiom Sensis (Siemens, Erlangen, Germany) by an independent operator not involved in the study or PCI procedure. QCA of the lesion, TIMI coronary flow, TIMI myocardial blush and TIMI frame count before and after PCI will be assessed.

Comprehensive echocardiogram with 2D-strain analysis will be done before and immediately after PCI procedure within 30 minutes after its end.

After the procedure, the patients who had an uneventful PCI will stay in the hospital for 24 h. Blood samples for Troponin I, creatin kinaze (CK) and CK-MB will be collected at 6, 12 and 24 h after the procedure, and for C reactive protein (CRP) after 24h. Complications of the interventions will be documented in the patients study file. Periprocedural myocardial necrosis is defined as rise in troponin I level three times 99th percentile upper limit of reference range, according to definition of myocardial infarction for clinical trials on coronary interventions.

After discharge from the hospital patients will be followed according to hospital protocol. Patients will be seen in an office visit 30 days and 6 months after baseline PCI procedure. At 12 months after baseline procedure patients' vital status will be assessed by telephone interview.

Statistical analysis

Continuous data will be summarized as the means ± SD. Categorical data will be summarized as counts and percentages. Unpaired t-tests will be used for comparing the continuous variables, if the distribution is normal, and Mann Whitney U test if the distribution is not normal. Chi-squared test and Fisher's exact test will be used for categorical vari¬ables. Multivariate logistic regression analysis will be performed to determine independent predictors of impaired IMR after PCI. Univariate analysis would be conducted first to identify potential factors for impaired IMR. The likelihood-ratio test will be used, and the variables with a p value < 0.2 would be included in the multivariate model. A p value of p<0.05 will be considered to be statistically significant. All statistical analyses will be performed with the PASWStatistics 18.0 statistical software (SPSS Inc, Chicago, Illinois, USA).

Based on the previous studies it was estimated that study sample size needed for expected difference in IMR values of 9 to be obtained between study groups (power 80%) is around 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* presence of the stable angina or positive stress test
* Canadian Cardiovascular Society (CCS) class less than IV
* single, de novo, native coronary artery lesion
* diameter stenosis greater than 70%.

Exclusion Criteria:

* left ventricular systolic function (LVEF) less than 30%
* acute coronary syndrome
* history of previous myocardial infarction in the territory supplied by the treated coronary artery
* existence of the collateral circulation to another coronary artery supplied by the treated vessel
* chronic total occlusion
* significant bifurcation lesion
* previous surgical revascularization
* significant renal function impairment (GFR less than 60ml/min) allergy to any constituents of trimetazidin, aspirin and antiplatelet medications used after PCI, contrast agents
* contraindication to adenosine use
* Parkinson disease
* parkinsonian symptoms, tremors, restless leg syndrome, and other related movement disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-04; Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
index of microcirculatory resistance | On day 2 during percutaneous coronary intervention
  Trimetazidine given on day 0 before elective percutaneous coronary intervention would decrease microvascular dysfunction by reducing index of microcirculatory resistance (IMR) measured by thermodilution method using coronary pressure and temperature wire on day 2 during PCI

SECONDARY OUTCOMES:
periprocedural myocardial necrosis | on day 2 after PCI
  Periprocedural myocardial necrosis will be measured by collecting blood samples for Troponin I, CK and CK-MB at 6, 12 and 24 h after the procedure.

OTHER OUTCOMES:
change in 2D myocardial strain | on day 2 30 minutes after completion of PCI procedure
  Comprehensive echocardiogram with 2D-strain analysis will be done before and immediately after PCI procedure to correlate change in IMR with possible change in 2D strain after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Petar Otasevic, MD, PhD, Study Director — Institute for cardiovascular diseases Dedinje Belgrade, Serbia
Locations (1):
- Institute for cardiovascular diseases Dedinje, Belgrade, Serbia

REFERENCES:
- [Background] Aussedat J, Ray A, Kay L, Verdys M, Harpey C, Rossi A. Improvement of long-term preservation of isolated arrested rat heart: beneficial effect of the antiischemic agent trimetazidine. J Cardiovasc Pharmacol. 1993 Jan;21(1):128-35. doi: 10.1097/00005344-199301000-00019. PMID 7678667
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Ng MK, Yeung AC, Fearon WF. Invasive assessment of the coronary microcirculation: superior reproducibility and less hemodynamic dependence of index of microcirculatory resistance compared with coronary flow reserve. Circulation. 2006 May 2;113(17):2054-61. doi: 10.1161/CIRCULATIONAHA.105.603522. Epub 2006 Apr 24. PMID 16636168
- [Background] Mangiacapra F, Peace AJ, Di Serafino L, Pyxaras SA, Bartunek J, Wyffels E, Heyndrickx GR, Wijns W, De Bruyne B, Barbato E. Intracoronary EnalaPrilat to Reduce MICROvascular Damage During Percutaneous Coronary Intervention (ProMicro) study. J Am Coll Cardiol. 2013 Feb 12;61(6):615-21. doi: 10.1016/j.jacc.2012.11.025. Epub 2013 Jan 2. PMID 23290547